CLINICAL TRIAL: NCT07288931
Title: A Comparative Study of Al18F-NOTA-LM3 Versus 68Ga-DOTATATE PET/CT for Tumor Detection in Patients With Pheochromocytoma and Paraganglioma
Brief Title: Al18F-NOTA-LM3 PET/CT in Patients With Pheochromocytoma and Paraganglioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALFLM3PPGL
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-01

CONDITIONS: Pheochromocytoma/Paraganglioma (PPGL)
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-LM3 and 68Ga-DOTATATE PET/CT scan (Experimental): Patients will perform an Al18F-NOTA-LM3 PET/CT as well as a 68Ga-DOTATATE PET/CT scan within one week, with a minimum 24-hour interval between scans.
  Interventions: Drug: Diagnostic Test: Al18F-NOTA-LM3; Drug: Diagnostic Test: 68Ga-DOTATATE

INTERVENTIONS:
Drug: Diagnostic Test: Al18F-NOTA-LM3 — Patients will receive a single intravenous injection of Al18F-NOTA-LM3. Subsequently, a PET/CT scan will be performed within 60 to 120 minutes post-injection.
Drug: Diagnostic Test: 68Ga-DOTATATE — Patients will receive a single intravenous injection of 68Ga-DOTATATE. Subsequently, a PET/CT scan will be performed within 40 to 60 minutes post-injection.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance of Al18F-NOTA-LM3 PET/CT and compare it with 68Ga-DOTATATE PET/CT in patients with pheochromocytoma/paraganglioma (PPGL).

DETAILED DESCRIPTION:
68Ga-based somatostatin receptor (SSTR) PET/CT has emerged as the cornerstone for staging and monitoring metastatic pheochromocytoma and paraganglioma (mPPGL), including its integral theranostic role in selecting patients for peptide receptor radionuclide therapy (PRRT). Compared to conventional 68Ga-DOTA-SSA analogs, 18F-labeled SSTR antagonists offer advantages including higher yield, superior image resolution, and longer half-life, potentially facilitating clinical workflow. Al18F-NOTA-LM3 is an SSTR2-specific antagonist developed as a PET tracer, with preliminary data supporting its safety, favorable biodistribution, and effective lesion targeting. This study aims to evaluate the diagnostic efficacy of Al18F-NOTA-LM3 PET/CT compared to 68Ga-DOTATATE PET/CT in a cohort of patients with PPGL.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* Suspected or confirmed PPGL patients.

Exclusion Criteria:

* Combined with other types of tumors.
* Severe liver or renal dysfunction (ALT/AST≥5 ULN, GFR<30ml/min).
* Pregnant or breast-feeding women.
* Inability to perform PET/CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Detection Rate | From study completion to 6 months after completion.
  Compare the number of tumor detected by Al18F-NOTA-LM3 PET/CT and 68Ga-DOTATATE PET/CT

SECONDARY OUTCOMES:
Standardized Uptake Value (SUV) of Tumor | From study completion to 6 months after completion.
  Compare the SUVmax of tumor derived from Al18F-NOTA-LM3 and 68Ga-DOTATATE PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China